CLINICAL TRIAL: NCT02766075
Title: A Supervised TAVR Exercise Program (STEP) for Patients Prior to Undergoing Transcatheter Aortic Valve Replacement (TAVR): A Pilot Study
Brief Title: A STEP for Patients Prior to Undergoing TAVR: A Pilot Study
Acronym: STEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: OSF Healthcare System (Other)
Collaborators: HeartCare Midwest (Unknown); University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 837484
Record Dates: First submitted 2016-04-28; First posted 2016-05-09 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-04

CONDITIONS: Frail Elderly; Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Disease; Supervised TAVR Exercise Program
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised TAVR Exercise Program (STEP) (Experimental): Subjects in the experimental arm will participate in an individualized 4-week STEP prior to undergoing TAVR. All subjects will undergo serial frailty assessments by a blinded research assistant at baseline, pre-TAVR, and 30-days post-TAVR.
  Interventions: Behavioral: Supervised TAVR Exercise Program
- Standard of Care (No Intervention): Subjects in the no intervention arm will proceed with their TAVR after a minimum 4 weeks without an exercise intervention. All subjects will undergo serial frailty assessments by a blinded research assistant at baseline, pre-TAVR, and 30-days post-TAVR.

INTERVENTIONS:
Behavioral: Supervised TAVR Exercise Program — Individualized exercise program designed and implemented by licensed physical therapy clinicians in three 60-minute sessions per week for four weeks. Upon randomization, subjects in the Intervention Group will undergo an initial Dynamic Gait & Balance Assessment by a licensed physical therapy clinician. The physical therapy clinician will use this assessment to design and implement an individualized STEP in three 60-minute sessions per week for four weeks. Subjects will proceed with their pre-TAVR testing in conjunction with the STEP sessions.
  Arms: Supervised TAVR Exercise Program (STEP)

SUMMARY:
The aim of this pilot study is to establish whether a Supervised TAVR Exercise Program (STEP) can safely improve the frailty status in patients with symptomatic severe aortic valve stenosis prior to undergoing transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
TAVR is an approved alternative therapy for patients with severe aortic valve stenosis who are deemed inoperable or high-risk for surgical aortic valve replacement (SAVR). Despite a very high procedural success rate (>95%), mortality rates after TAVR at 1- and 2-year follow-up remain ≥25% and ≥34%, respectively. It is becoming increasingly evident that frailty, as a clinical syndrome, has a large impact on this long term mortality. In a study by Green, et al. frailty status was independently associated with increased 1-year mortality (OR=3.5) after TAVR. The investigators' own retrospective analysis showed that impaired mobility and malnutrition were significantly associated with a longer hospital length of stay (5 days vs. 3 days), and increased total cost (on average, an additional $10,000 per patient). Given the phenotype of frailty is characterized by reductions in muscle mass, strength, endurance and activity level, a STEP is ideally suited to counteract these impairments. This pilot study aims to establish whether a STEP can safely improve the frailty score in patients with symptomatic severe aortic valve stenosis prior to undergoing TAVR.

This single-center pilot study will be conducted in partnership between Heart Care Midwest (HCMW), OSF St. Francis Medical Center (OSF SFMC), and University of Illinois College of Medicine at Peoria (UICOMP). UICOMP Center of Outcomes Research will provide analytical support. The study will be funded by an operational research grant from OSF SFMC.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled to undergo first-time elective TAVR

Exclusion Criteria:

* Vulnerable populations including prisoners, pregnant females and patients less than 18 years age.
* Patients with history of unstable angina, myocardial infarction, or decompensated heart failure in the week prior to screening
* Patients with physical limitations (i.e. debilitating stroke, amputation, unable to complete initial screening frailty profile)
* Patients with advanced dementia or cognitive deficits (i.e. unable to follow instructions of initial screening frailty profile)
* Exercise-induced arrhythmias

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Frailty Score from Baseline to post-STEP | Baseline, 6-weeks

SECONDARY OUTCOMES:
Adverse Events | 6-weeks
Change in Frailty Score from Baseline to 30-days post-TAVR | Baseline, 30-days post-TAVR
Change in Gait Speed (5-Meter Walk Test) from Baseline to post-STEP | Baseline, 6-weeks
Change in Gait Speed (5-Meter Walk Test) from Baseline to 30-days post-TAVR | Baseline, 30-days post-TAVR
Change in Grip Strength (Dynamometer) from Baseline to post-STEP | Baseline, 6-weeks
Change in Grip Strength (Dynamometer) from Baseline to 30-days post-TAVR | Baseline, 30-days post-TAVR
Change in Independent Activity (Katz Activities of Daily Living Survey) from Baseline to post-STEP | Baseline, 6-weeks
Change in Independent Activity (Katz Activities of Daily Living Survey) from Baseline to to 30-days post-TAVR | Baseline, 30-days post-TAVR
Change in Malnutrition (Serum Albumin Level) from Baseline to 30-days post-TAVR | Baseline, 30-days post-TAVR

CONTACTS AND LOCATIONS:
Overall Officials: Jay N Patel, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF St. Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No